CLINICAL TRIAL: NCT02385136
Title: Temozolomide and Concomitant Whole Brain Radiotherapy in NSCLC Patients With Brain Metastases: A Randomized Trial
Brief Title: Temozolomide and Concomitant Whole Brain Radiotherapy in NSCLC Patients With Brain Metastases
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Hangzhou Cancer Hospital (Other)
Responsible Party: Principal Investigator, chenjianxiang, Dr Chen, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: zjzlyy 2015-1-5
Record Dates: First submitted 2015-03-03; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: NSCLC
Keywords: NSCLC; Radiotherpy; Temozolomide
MeSH Terms: interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WBRT plus TMZ arm (Experimental): whole brain radiotherapy (WBRT) concomitantly with temozolomide (TMZ)
  Interventions: Drug: Temozolomide
- WBRT (No Intervention): whole brain radiotherapy (WBRT)

INTERVENTIONS:
Drug: Temozolomide
  Arms: WBRT plus TMZ arm

SUMMARY:
The purpose of this study is to evaluate the safety profile and efficacy of whole brain radiotherapy (WBRT) concomitantly with temozolomide (TMZ) in patients with brain metastases (BM).Patients with BM were randomly assigned to 30 Gy of WBRT with or without concomitant TMZ (75 mg/m2/d) plus two cycles of TMZ (200 mg/m2/d for 5 days).

ELIGIBILITY:
Inclusion Criteria:

* histologically diagnosed as NSCLC, stage IVb [ (American Joint of Cancer Committee(AJCC), 2002) ], Brain metastasis
* no history of hypertension or diabetes.

Exclusion Criteria:

* the brain tumor diameter >5cm; RPA class =3; pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 1 month post procedure
Time to central nervous system progress which was confirmed by MRI | 1 to 24 months post procedure

SECONDARY OUTCOMES:
The Quality of Life | 0 to 24 months post procedure
Overall Survival | 1 to 24 months post procedure
Toxicity as measured by CTCAE V4.0 | 0 to 24 months post procedure